CLINICAL TRIAL: NCT02013843
Title: Treatment of Overweight and Obese Children - the "Holbaek-Method" in a Municipality Based Treatment Program.
Brief Title: Treatment of Overweight and Obese Children -Using the "Holbaek-Method" in a Municipality Based Treatment Program.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Pernille Maria Mollerup, MD, Holbaek Sygehus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TCOCmunicipalities; Region Sjaelland 2012 (Other Grant/Funding Number: Region Sjaelland)
Record Dates: First submitted 2013-12-06; First posted 2013-12-17 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Pediatric Obesity; Dyslipidemia; Hypertension; Diabetes; Quality of Life
Keywords: Pediatric obesity; Community-based treatment; dyslipidemia; hypertension; diabetes
MeSH Terms: conditions — Pediatric Obesity; Dyslipidemias; Hypertension; Diabetes Mellitus | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Community-based treatment (Other): Overweight and obese children are seen on a regular basis by health care professionals in the 8 communities included in the project. The care providers are all trained thoroughly in using the "Holbaek-method" for treatment of pediatric obesity.
  Interventions: Behavioral: Community-based treatment of overweight and obesity

INTERVENTIONS:
Behavioral: Community-based treatment of overweight and obesity — Community based treatment of overweight and obese children using the "Holbaek-method".

SUMMARY:
In the present study the effect of a community-based treatment of overweight and obese children is analyzed. The treatment-method is based on the principals and the method used in the Children Obesity Clinic in the Pediatric department i Holbaek. The effect is evaluated by the change in body mass index standard deviation score, change in blood pressure standard deviation score, quality of life and concentration of fasting blood lipids and glucose during one year of treatment.

DETAILED DESCRIPTION:
In the present study the effect of a community-based treatment of overweight and obese children is analyzed. The treatment-method is based on the principals and the method used in the Children Obesity Clinic in the Pediatric department i Holbaek and the care providers in each of the eight municipalities included are thought thoroughly to use this method.

The treatment effect is evaluated after one year, and the effect is assessed by the change in body mass index standard deviation score, change in blood pressure standard deviation score, quality of life (PedsQL), body composition and concentration of fasting blood lipids and glucose.

ELIGIBILITY:
Inclusion Criteria:

- Body mass index above 90-percentile for age and gender

Exclusion Criteria:

* None

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1007 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Body mass index standard deviation score | 1 year
  primary outcome is the change in body mass index standard deviation score during 12 month treatment of overweight and obesity.

SECONDARY OUTCOMES:
Change in blood pressure standard deviation score | 1 year
Change in the concentration of blood lipids | 1 year
change in the concentration of fasting blood-glucose, HBA1C and insulin | 1 year
Change in body composition measured by Tanita BC 418 | 1 year
Change in quality of life assessed by PedsQL | 1 year

OTHER OUTCOMES:
cost effectiveness | 1 year
  Assessed by the amount of hours used per child per year in each municipality

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric department, Holbæk, Denmark

REFERENCES:
- [Background] Holm JC, Gamborg M, Neland M, Ward L, Gammeltoft S, Heitmann BL, Sorensen TI, Ibsen KK. Longitudinal changes in blood pressure during weight loss and regain of weight in obese boys and girls. J Hypertens. 2012 Feb;30(2):368-74. doi: 10.1097/HJH.0b013e32834e4a87. PMID 22157326
- [Background] Holm JC, Gamborg M, Bille DS, Gr Nb K HN, Ward LC, Faerk J. Chronic care treatment of obese children and adolescents. Int J Pediatr Obes. 2011 Aug;6(3-4):188-96. doi: 10.3109/17477166.2011.575157. Epub 2011 May 2. PMID 21529264
- [Derived] Mollerup PM, Nielsen TRH, Bojsoe C, Kloppenborg JT, Baker JL, Holm JC. Quality of life improves in children and adolescents during a community-based overweight and obesity treatment. Qual Life Res. 2017 Jun;26(6):1597-1608. doi: 10.1007/s11136-017-1504-x. Epub 2017 Feb 17. PMID 28213684